CLINICAL TRIAL: NCT00487929
Title: Phase 4 Study of the Relationship Between the Oxidative Stress and the Development of Cardiovascular Complications in the Sleep Apnea-hypopnea Syndrome (SAHS). Effect of the Treatment With CPAP
Brief Title: Oxidative Stress and Cardiovascular Morbidity in Sleep Apnea-Hypopnea Syndrome (SAHS)
Acronym: OSCAMSA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Universitario La Paz (Other)
Responsible Party: Francisco Garcia-Rio, Hospital Universitario La Paz
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: HULP051937
Record Dates: First submitted 2007-06-18; First posted 2007-06-19 (Estimated); Last update posted 2013-04-02 (Estimated); Status verified 2008-10

CONDITIONS: Sleep Apnea; Cardiovascular Diseases
Keywords: sleep apnea; morbidity; cardiovascular; cpap; oxidative stress
MeSH Terms: conditions — Sleep Apnea Syndromes; Cardiovascular Diseases; Microcephaly, Primary Autosomal Recessive, 6

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CPAP (Experimental): Continuous positive airway pressure
  Interventions: Device: nasal CPAP
- Sham CPAP (Sham Comparator): Sham nasal continuous positive airway pressure
  Interventions: Device: Sham CPAP

INTERVENTIONS:
Device: nasal CPAP — Nocturnal
  Arms: CPAP
Device: Sham CPAP — Nocturnal
  Arms: Sham CPAP

SUMMARY:
The purpose of this study is to compare the levels of 8-isoprostane and other oxidative stress biomarkers in plasma and condensed exhaled air between patients with SAHS and cardiovascular complications, patients with SAHS without cardiovascular complications and control subjects. To evaluate the effect of three months of treatment with CPAP on the oxidative stress biomarkers.

DETAILED DESCRIPTION:
Aim: To compare the levels of 8-isoprostane and other oxidative stress biomarkers in plasma and condensed exhaled air between patients with SAHS and cardiovascular complications, patients with SAHS without cardiovascular complications and control subjects. To evaluate the effect of three months of treatment with CPAP on the oxidative stress biomarkers.

Design: randomized, double blind, of parallel groups and controlled with placebo study.

Study subjects: 53 patients with SAHS (23 with cardiovascular complications and 30 without cardiovascular complications), 23 patients with cardiovascular diseases without SAHS and 23 control subjects.

Interventions: Three months of treatment with therapeutic CPAP or with sham CPAP (placebo).

Determinations: clinical (cardiovascular morbidity) and anthropometric data. Fat free corporal mass, echocardiography, spirometry, ambulatory monitoring of the arterial pressure, endothelial reactivity. Oxidative stress biomarkers (8-isoprostane, homocysteine, HIF-1, NFkB, AP-1, VEGF, ET-1, TNF-alpha, IL-1, IL-6, ICAM-1, VCAM-1, nitrates and nitrites) in plasma and condensed exhaled air.Peripheral sensitivity to hypoxia. Urinary excretion of catecholamines.

ELIGIBILITY:
Inclusion Criteria:

* Sleep apnea-hypopnea syndrome (AHI > 5)
* Excessive sleepiness (ESS > 11)
* No previous CPAP treatment

Exclusion Criteria:

* Blood pressure > 180/120 mmHg.
* Secondary hypertension
* Professional driver
* COPD, asthma, bronchiectasis, lung cancer, restrictive lung disorder, chest wall disease
* Neuromuscular disease or thyroid function abnormalities
* Morbid obesity (BMI > 40 Kg/m2).
* Respiratory infection in the 2 last months.
* Anemia (Hb < 10 g/dl) or polyglobulia (Hct > 55%).
* Diurnal hypercapnia (PaCO2 > 45 mmHg) or moderate hypoxemia (PaO2 < 70 mmHg).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-06; Primary Completion 2012-04 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Plasmatic 8-isoprostane concentration | three months

SECONDARY OUTCOMES:
Plasmatic and condensed exhaled air concentrations of homocysteine, HIF-1, NFkB, AP-1, VEGF, ET-1, TNF-alpha, IL-1, IL-6, ICAM-1, VCAM-1, nitrates and nitrites. | three months

CONTACTS AND LOCATIONS:
Overall Officials: Francisco García-Rio, PhD, Study Chair — Servicio de Neumología. Hospital Universitario La Paz
Locations (1):
- Hospital Universitario La Paz, Madrid, Madrid, Spain